CLINICAL TRIAL: NCT06356727
Title: Microvascular Dysfunction Assessment to Predict Left Ventricular Reverse Remodeling in Idiopathic Dilated Cardiomyopathy
Brief Title: Microvascular Dysfunction Assessment to Predict Left Ventricular Reverse Remodeling
Acronym: MICROREV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Roberto Scarsini, Principal investigator, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 121CET-MICROREV-DCM
Record Dates: First submitted 2024-03-30; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Heart Failure; Left Ventricular Dysfunction; Idiopathic Dilated Cardiomyopathy
Keywords: coronary microvascular dysfunction; heart failure; left ventricular reverse remodeling; optimal medical therapy
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Cardiomyopathy, Dilated

STUDY DESIGN:
Intervention Model Description: Prospective multicenter single-arm experimental study. The study aims to perform a functional study of the coronary microcirculation with pressure guides, in patients with new diagnoses of dilated cardiomyopathy and clinical indication for coronary angiography. Following this, a multiparametric imaging study with transthoracic echo cardiography will be performed. 12 months after the optimization of medical therapy, the patient will receive a clinical, laboratory and instrumental re-evaluation of transthoracic cardiac color Doppler. The primary endpoint is the recovery of left ventricular function on cardiac imaging. Follow up will continue up to 5 years from enrollment through telephone contacts, outpatient visits and review of clinical data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microvascular assessment (Experimental): Coronary microvascular assessment
  Interventions: Diagnostic Test: Thermodilution based assessment of coronary microcirculation

INTERVENTIONS:
Diagnostic Test: Thermodilution based assessment of coronary microcirculation — Coronary microvascular assessment with the derivation of CFR, IMR and MRR will be performed using a standard pressure/thermodilution guidewire.

SUMMARY:
Patients presenting with idiopathic dilated cardiomyopathy and left ventricle dysfunction (LVEF <40%), naive of anti-remodeling cardiac medical therapy, will undergo invasive coronary microvascular assessment based on thermodilution. The primary endpoint, namely the left ventricle reverse remodeling, will be assessed after 12 months of optimal medical therapy based on transthoracic echocardiography. The primary endpoint will be evaluated by an independent central core lab. Patients enrolled in the study will be followed for a period of 5 years to monitor their clinical status. During the study period participants may undergo multimodality diagnostic tests including ECG telemetry monitoring, cardiopulmonary exercise testing, cardiovascular cardiac magnetic resonance.

DETAILED DESCRIPTION:
This is a prospective, multicentric, single-arm explorative clinical study in patients presenting with heart failure and idiopathic dilated cardiomyopathy with LVEF ≤ 40%. Patients identified as eligible for the protocol will be asked for written informed consent to participate in the study.

After appropriate treatment of the acute heart failure phase, participants will undergo coronary angiography to rule out obstructive coronary disease.

Fractional flow reserve (FFR) will be assessed as per standard clinical practice and a value ≤ 0.80 will be considered abnormal. Microvascular assessment will be performed using the same pressure/thermodilution guidewire used for FFR assessment with the derivation of coronary flow reserve (CFR), index of microcirculatory resistance (IMR) and the microvascular resistance reserve (MRR).

Steady-state hyperemia will be obtained using an intravenous adenosine infusion or intracoronary papaverine as per routine clinical practice.

The primary endpoint will be assessed based on the variation of echocardiographic indices from the baseline to 12-month follow up. Transthoracic echocardiography will be performed to confirm the diagnosis and obtain information about adverse cardiac remodeling and after 12 months of optimal medical therapy to evaluate reverse remodeling.

Patients will be clinically managed by a dedicated heart failure team to optimize medical therapy and organize the follow-up.

Patients enrolled in the study will be clinically followed for a period of 5 years to monitor the clinical status and report major adverse cardiac events.

During the study period participants may undergo multimodality diagnostic tests according to the recent international guidelines. Data from these tests will be collected if the test will be performed per clinical practice:

1. 3-leads ECG telemetry monitoring (or 24 hours Holter ECG) to detect or quantify atrial and/or ventricular arrhythmias during the hospitalization.
2. N-terminal pro-B-type natriuretic peptide (NT - proBNP).
3. Cardiopulmonary exercise testing (CPET) to assess functional capacity.
4. Contrast enhanced cardiac magnetic resonance. CMR assessment may be repeated at 12 months follow-up.
5. Genetic counseling and genetic testing, performed by an appropriately trained healthcare professional is recommended in patients with idiopathic DCM by the latest international guidelines to enable diagnosis, prognostication, therapeutic stratification.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged >18 years
* First diagnosis of idiopathic DCM (defined according to the most recent ESC Guidelines) with LVEF ≤ 40% and clinical indication to diagnostic coronary angiography
* Willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Obstructive CAD (defined as angiographically intermediate disease [50%-70%] with impaired FFR or as angiographically severe disease [>70%] in 1 or more epicardial vessels)
* History of previous myocardial infarction, percutaneous revascularization or coronary-aortic bypass graft (CABG) surgery
* Valvular heart disease (rheumatic heart disease, severe aortic stenosis, severe aortic regurgitation, severe primary mitral regurgitation)
* Infective endocarditis
* Congenital heart disease
* Peripartum cardiomyopathy
* Acute myocarditis (detected by endomyocardial biopsy - histological criteria - or by CMR - Lake Louis criteria) and pericarditis
* Persistent tachyarrhythmias (documented persistent high-rate supraventricular arrhythmias)
* Excessive alcohol intake (>80 g/die for at least five years)
* History of chemotherapy (anthracycline therapy, cumulative dosages >250 mg/m2)
* History of uncontrolled arterial hypertension (blood pressure >160/100 mmHg)
* Stage IV and V of chronic kidney disease (eGFR < 30 ml/min, estimated through CKD - EPI Creatinine Equation)
* Allergy or other contraindication to iodinated contrast and/or adenosine
* Chronic resting O2 saturation <85%
* Pregnancy or suspected pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Left ventricular reverse remodeling (LVRR) | After 12 months of guidelines directed optimal medical therapy
  LVRR, defined as LVEF increase ≥ 10% and LVEDDi decrease ≥ 10%, will be assessed with transthoracic echocardiography and analyzed off-line by an independent central corelab.

SECONDARY OUTCOMES:
Adverse clinical events | Up to 5 years
  Composite of cardiovascular death, new hospitalization for HF, ICD implantation, heart transplantation or ventricular mechanical assistance implantation during follow-up in patients with and without coronary microvascular dysfunction
Rate of LVRR at cardiac magnetic resonance | After 12 months of guidelines directed OMT
  LVRR, defined as LVEF increase ≥ 10% and LVEDDi decrease ≥ 10%, in patients who will undergo CMR at baseline and at 12 months follow up.
Changes in functional capacity at cardiopulmonary exercise test | After 12 months of guidelines-defined OMT
  Variations of VO2 max at CPET after 12 months of guidelines-defined OMT
Prevalence of different CMD endotypes and their correlation with the severity of adverse cardiac remodeling. | At baseline
  CMD endotypes (defined as IMR >25 units and/or CFR <2)
Left ventricle adverse cardiac remodeling at cardiovascular magnetic resonance. | At baseline
  Measures of LV adverse remodeling at CMR

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Scarsini, MD PhD, Principal Investigator — Azienda Ospedaliera Universitaria di Verona
Locations (9):
- Italy (9):
  - Azienda Ospedaliera Universitaria di Ferrara, Ferrara
  - Cardiothoracic and Vascular Department (DICATOV) IRCCS, Ospedale Policlinico San Martino, Genova
  - Istituto di Ricovero e Cura a Carattere Scientifico (IRCCS) dell'Ospedale San Raffaele, Milan
  - Ospedale Galeazzi di Sant'Ambrogio IRCCS, Milan
  - University of Naples Federico II, Naples
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Rome
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
  - Azienda Ospedaliera Universitaria di Verona, Verona

IPD SHARING:
Plan to Share IPD: Yes
Yes.
Supporting Information: Study Protocol
Time Frame: The present study is powered for assessing left ventricular reverse remodeling in patients with and without coronary microvascular dysfunction. However, the study is not powered for clinical adverse events. In order to obtain compelling evidence on this latter endpoint, the data of the present study will be merged with those of clinical studies sharing the same inclusion and exclusion criteria and study interventions.
  Data will be available for individual patient level analysis in order to merge our data with other studies sharing inclusion and exclusion criteria. Data will be available after the completion of the primary endpoint.
Access Criteria: Direct request to study Principal Investigator.

REFERENCES:
- [Background] Arbelo E, Protonotarios A, Gimeno JR, Arbustini E, Barriales-Villa R, Basso C, Bezzina CR, Biagini E, Blom NA, de Boer RA, De Winter T, Elliott PM, Flather M, Garcia-Pavia P, Haugaa KH, Ingles J, Jurcut RO, Klaassen S, Limongelli G, Loeys B, Mogensen J, Olivotto I, Pantazis A, Sharma S, Van Tintelen JP, Ware JS, Kaski JP; ESC Scientific Document Group. 2023 ESC Guidelines for the management of cardiomyopathies. Eur Heart J. 2023 Oct 1;44(37):3503-3626. doi: 10.1093/eurheartj/ehad194. No abstract available. PMID 37622657
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Merlo M, Pyxaras SA, Pinamonti B, Barbati G, Di Lenarda A, Sinagra G. Prevalence and prognostic significance of left ventricular reverse remodeling in dilated cardiomyopathy receiving tailored medical treatment. J Am Coll Cardiol. 2011 Mar 29;57(13):1468-76. doi: 10.1016/j.jacc.2010.11.030. PMID 21435516
- [Background] Rosano GMC, Moura B, Metra M, Bohm M, Bauersachs J, Ben Gal T, Adamopoulos S, Abdelhamid M, Bistola V, Celutkiene J, Chioncel O, Farmakis D, Ferrari R, Filippatos G, Hill L, Jankowska EA, Jaarsma T, Jhund P, Lainscak M, Lopatin Y, Lund LH, Milicic D, Mullens W, Pinto F, Ponikowski P, Savarese G, Thum T, Volterrani M, Anker SD, Seferovic PM, Coats AJS. Patient profiling in heart failure for tailoring medical therapy. A consensus document of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2021 Jun;23(6):872-881. doi: 10.1002/ejhf.2206. Epub 2021 May 20. PMID 33932268
- [Background] Del Buono MG, Montone RA, Camilli M, Carbone S, Narula J, Lavie CJ, Niccoli G, Crea F. Coronary Microvascular Dysfunction Across the Spectrum of Cardiovascular Diseases: JACC State-of-the-Art Review. J Am Coll Cardiol. 2021 Sep 28;78(13):1352-1371. doi: 10.1016/j.jacc.2021.07.042. PMID 34556322
- [Background] Gulati A, Ismail TF, Ali A, Hsu LY, Goncalves C, Ismail NA, Krishnathasan K, Davendralingam N, Ferreira P, Halliday BP, Jones DA, Wage R, Newsome S, Gatehouse P, Firmin D, Jabbour A, Assomull RG, Mathur A, Pennell DJ, Arai AE, Prasad SK. Microvascular Dysfunction in Dilated Cardiomyopathy: A Quantitative Stress Perfusion Cardiovascular Magnetic Resonance Study. JACC Cardiovasc Imaging. 2019 Aug;12(8 Pt 2):1699-1708. doi: 10.1016/j.jcmg.2018.10.032. Epub 2019 Jan 16. PMID 30660522